CLINICAL TRIAL: NCT03983291
Title: Facial Rehabilitation of Wellbeing in Depression: a Randomized Controled Trial of a Facial Physiotherapeutic Exercise Program in the Treatment of Depression
Brief Title: FaReWell Depression - Facial Exercise Program to Treat Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zentrum für Angst und Depressionsbehandlung Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 1.1
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: For six weeks one arm receives the FaReWell Depression intervention and one arm receives a control resting intervention. The former arm continues on the FaReWell Depression intervention while the latter arm is switched to the FaReWell Depression intervention for another six weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FaReWell Depression (Experimental): Physiotherapeutic exercises for the relaxation of facial muscles associated with the expression of negative emotions and for the activation and strengthening of facial muscles associated with the expression of positive emotions 15 minutes daily
  Interventions: Behavioral: FaReWell Depression
- Resting exercise (Placebo Comparator): Resting 15 minutes daily
  Interventions: Behavioral: FaReWell Depression

INTERVENTIONS:
Behavioral: FaReWell Depression — Facial massage and force exercise

SUMMARY:
This study investigates if a physiotherapeutic exercise program designed to relax facial muscles associated with the expression of negative emotions and to activate and strengthen facial muscles associated with the expression of positive emotions can reduce the symptoms of depression and improve wellbeing and quality of life in the affected patients.

DETAILED DESCRIPTION:
Activity of the facial musculature expresses emotions, but also generates proprioceptive signals to the emotional brain that maintain and reinforce the expressed emotions. This has been described by Charles Darwin and William James in the facial feedback hypothesis.

Studies have shown that interruption of facial feedback by the injection of botulinum toxin into the corrugator and procerus muscles, which express negative emotions like sadness, anger, and fear, can reduce the symptoms of depression.

In the present study we investigate, if similar effects can be achieved by a relaxing massage of these and other muscles that are associated with the expression of negative emotions and if strengthening exercises of muscles that express positive emotions, the zygomaticus and orbicularis oculi muscles, can contribute to the rehabilitation of positive emotionality in depression. After instruction by a physiotherapist, participants will practice the exercises daily for 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate unipolar depression
* Stable treatment for at least 6 weeks

Exclusion Criteria:

* Organic mental disorders
* Mental disorders due to psychoactive substance use
* Schizophrenia and other psychotic disorders
* Previous cosmetic procedures (botulinum toxin, fillers, lifting)
* Facial palsy
* Facial skin disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | 6 weeks
  The Montgomery-Asberg Depression Rating Scale (MADRS) is an expert rating scale with 10 items for the measurement of the severity of depressive symptoms. Change in depression severity is measured as change in the total score of the scale (0-60 points).

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | 3, 9, 12 weeks
  The Montgomery-Asberg Depression Rating Scale (MADRS) is an expert rating scale with 10 items for the measurement of the severity of depressive symptoms. Change in depression severity is measured as change in the total score of the scale (0-60 points).
Change in Patient-Health-Questionnaire-9 (PHQ-9) | 3, 6, 9, 12 weeks
  The Patient-Health-Questionnaire-9 (PHQ-9) is a self-rating scale with 9 items for the measurement of the severity of depressive symptoms. Change in depression severity is measured as change in the total score of the scale (0-27 points).
Change in Snaith-Hamilton-Pleasure-Scale (SHAPS-D) | 3, 6, 9, 12 weeks
  The Snaith-Hamilton-Pleasure-Scale (SHAPS-D) is a self-rating scale with 14 items for the measurement of pleasure. Change in anhedonia (inability to experience pleasure) is measured as change in the total score of the scale (0-14 points).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Waldvogel, PhD, Principal Investigator — Zentrum für Angst und Depressionsbehandlung Zürich
Locations (1):
- Zentrum für Angst- und Depressionsbehandlung, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No